CLINICAL TRIAL: NCT02673164
Title: Stem Cell Therapy in IschEmic Non-treatable Cardiac Disease - SCIENCE A European Multi-Centre Trial
Brief Title: Stem Cell Therapy in IschEmic Non-treatable Cardiac Disease
Acronym: SCIENCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: JKastrup (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor-Investigator, JKastrup, MD Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCIENCE
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Heart Failure
Keywords: Heart failure; stem cell; adipose derived stem cell; Stem cell therapy; ischemic heart disease
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSCC_ASC (Active Comparator): Cardiology Stem Cell Centre_adipose derived stem cells (CSCC_ASC)
  Interventions: Biological: CSCC_ASC
- Placebo (Placebo Comparator): Saline
  Interventions: Biological: CSCC_ASC

INTERVENTIONS:
Biological: CSCC_ASC — The stem cells will be injected directly into the myocardium using the NOGA XP system (BDS, US)
  Other Names: Cardiology Stem Cell Centre_adipose derived stem cells

SUMMARY:
The aim of the SCIENCE study is, in an international multicentre double-blind placebo-controlled study, to investigate efficacy of direct intra-myocardial injection of 100 mio. allogeneic Cardiology Stem Cell Centre_adipose derived stem cells (CSCC_ASCs) in patients with reduced left ventricular Ejection Fraction (EF) (≤45%) and heart failure.

DETAILED DESCRIPTION:
The aim of the SCIENCE study is, in an international multicentre double-blind placebo-controlled study, to investigate efficacy of direct intra-myocardial injection of 100 mio. allogeneic Cardiology Stem Cell Centre_adipose derived stem cells (CSCC_ASCs) in patients with reduced left ventricular EF (≤45%) and heart failure.

The primary objective is to investigate the regenerative capacity of direct intra-myocardial injection of 100 mio. allogeneic CSCC_ASCs in patients with reduced left ventricular EF (≤45%) and heart failure in a double-blind placebo-controlled design.

A total of 138 patients with will be enrolled in the study and treated in a 2:1 randomization with either CSCC_ASC or placebo (saline).

ELIGIBILITY:
Inclusion Criteria:

1. 30 to 80 years of age
2. Signed informed consent
3. Chronic stable ischemic heart disease
4. Symptomatic heart failure New York Heart Association (NYHA) class II-III
5. EF ≤ 45% on echocardiography, Computerized Tomography (CT) or Magnetic Resonances Imaging (MRI) scan
6. Plasma NT-pro-BNP > 300 pg/ml (> 35 pmol/L)
7. Maximal tolerable heart failure medication
8. Heart failure medication unchanged two months prior to inclusion. Changes in diuretics accepted.
9. No option for percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG)
10. Patients who have had PCI or CABG within six months of inclusion must have a new coronary angiography less than one month before inclusion or at least four months after the intervention to rule out early restenosis
11. Patients cannot be included until three months after implantation of a cardiac resynchronisation therapy device (CRTD) and until 1 month after an ICD unit

Exclusion Criteria:

1. Heart Failure (NYHA class I or IV)
2. Acute coronary syndrome with acute reversible elevation of CKMB or troponins, stroke or transitory cerebral ischemia within six weeks of inclusion. Constant elevated troponin due to renal failure, heart failure etc. do not exclude the patient.
3. Other revascularisation treatment within four months of treatment
4. If clinically indicated the patient should have a coronary angiography before inclusion
5. Moderate to severe aortic stenosis (valve area < 1.3 cm2) or valvular disease with option for surgery or interventional therapy.
6. Aortic valve replacement with an artificial heart valve. However, a trans-septal treatment approach can be considered in these patients.
7. If the patient is expected to be candidate for MitraClip therapy of mitral regurgitation in the 12 months follow-up period.
8. Diminished functional capacity for other reasons such as: obstructive pulmonary disease (COPD) with forced expiratory volume (FEV) <1 L/min, moderate to severe claudication or morbid obesity
9. Clinical significant anaemia (haemoglobin < 6 mmol/L), leukopenia (leucocytes < 2 109/L), leucocytosis (leucocytes > 14 109/L) or thrombocytopenia (thrombocytes < 50 109/L)
10. Reduced kidney function (estimated Glomerular Filtration Rate (eGFR) < 30 ml/min)
11. Left ventricular thrombus
12. Anticoagulation treatment that cannot be paused during cell injections. Patients can continue with platelet inhibitor treatment
13. Patients with reduced immune response or known anti-HLA (human leukocyte antigen) antibodies
14. History with malignant disease within five years of inclusion or suspected malignity - except treated skin cancer other than melanoma
15. Pregnant women
16. Other experimental treatment within four weeks of baseline tests
17. Participation in another intervention trial
18. Life expectancy less than one year
19. Known hypersensitivity to Dimethyl sulfoxide (DMSO), penicillin and streptomycin

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
left ventricle end-systolic volume (LVESV) | 6 months
  The primary endpoint is change in left ventricle end-systolic volume (LVESV) from baseline to 6 months follow-up measured by ECHO, MR and CT between CSCC_ASC and placebo treated

SECONDARY OUTCOMES:
Safety - Serious adverse events | 6 months
  Incidence and severity of serious adverse events and suspected unrelated serious adverse events 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, Professor MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- 2014 Department of Cardiology, The Heart Centre, University Hospital Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared for Scientific collaboration